CLINICAL TRIAL: NCT02341586
Title: A Randomized Control Trial of the Lucky Iron Fish to Improve Hemoglobin Concentration in Women in Preah Vihear, Cambodia
Brief Title: Lucky Iron Fish Home Fortification of Iron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: NCHADS - Ministry of Health of Cambodia (Other); University of Guelph (Other)
Responsible Party: Principal Investigator, Tim Green, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H14-02551
Record Dates: First submitted 2015-01-09; First posted 2015-01-19 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Anemia; Anemia, Iron-Deficiency; Hemoglobinopathies
Keywords: Malaria; Cambodia; Iron; Childbearing Age; Women; Home Fortification
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency; Hemoglobinopathies; Malaria | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lucky Iron Fish (Experimental): This group will receive a Lucky Iron Fish to use during cooking.
  Interventions: Other: Lucky Iron Fish - home fortification system
- 18 mg iron (Active Comparator): This group will receive a daily oral iron supplement.
  Interventions: Dietary Supplement: 18 mg elemental iron
- Control group (Other): This group will receive nutrition education
  Interventions: Other: Nutrition Education

INTERVENTIONS:
Other: Lucky Iron Fish - home fortification system — The Lucky Iron Fish (LIF) is an ingot used during cooking as an in-home fortification system of iron. The LIF works on the same principle as cast iron pots and pans by increasing dietary intake of iron but is small and lightweight. The LIF was designed in collaboration with village elders and community members to ensure it would be accepted in Cambodia. The iron ingot resembles a local fish believed to be lucky among villages in Cambodia, contributing to the acceptability of the ingot.
  Arms: Lucky Iron Fish
Dietary Supplement: 18 mg elemental iron — This dose of iron is the recommend dietary allowance (RDA) for iron for this cohort. Women will receive one-on-one instructions on how best to consume their tablet (for example, with food).
  Arms: 18 mg iron
Other: Nutrition Education — This group will receive education containing key messages around anemia, malaria, iron intake, and dietary diversity.
  Arms: Control group

SUMMARY:
The purpose of this research is to determine if cooking with an iron ingot called the Lucky Iron Fish (LIF) increases the hemoglobin status in women of childbearing age living in Preah Vihear, Cambodia. The investigators hypothesize that the use of the LIF during cooking over a 12-month period will be as efficacious at increasing hemoglobin concentration as iron supplements (18 mg elemental iron) and will be more efficacious than the control.

DETAILED DESCRIPTION:
Background: Anemia is prevalent in Cambodia, affecting ~44% of women. The causes of anemia are multifactorial. Globally, the most common form is iron deficiency anemia (IDA), which can lead to adverse perinatal health outcomes. In Cambodia, there is evidence that suggests hemoglobinopathies (genetic hemoglobin [Hb] disorders) are prevalent (~50%) and are a major contributor to anemia. In Preah Vihear province, Cambodia, the estimated prevalence of malaria is ~12.3%. Malaria contributes to anemia through a decrease in the production of red blood cells, and an increased destruction of red blood cells.

In Cambodia, iron supplements are recommended to treat anemia, however there is evidence of low compliance among women. The use of cast iron pots has proven to be an effective alternative to prevent and reduce IDA in developing countries. However, cast iron pots are not commonly used in Cambodia because they are expensive, difficult to clean, and heavy. A novel alternative is the Lucky Iron Fish (LIF), which is an iron ingot used during cooking as an in-home fortification system of iron transfer. The LIF ingot is small, lightweight, and easy to clean. Previous research in Cambodia confirmed the acceptance of the LIF to be high, but findings from this study were inconclusive and had several limitations.

Objective: The primary objective of this study is to determine the efficacy of the LIF to increase Hb concentration in Cambodian women of reproductive age.

Methods: A total of 330 women (18-49 y) with mild or moderate anemia (Hb 80-120 g/L) from rural Preah Vihear, Cambodia will be recruited to one of three arms to receive LIF, 18 mg elemental iron, or a placebo. Women with severe anemia will be excluded and referred for treatment. All three groups will receive nutrition education. Monitoring will be conducted monthly to measure compliance.

A trained, Khmer-speaking interviewer will meet with the women to explain the details of the study as per the consent form. Once consent is obtained the trained interviewer will measure hemoglobin status using a hemocue device to confirm eligibility of the study. If eligible, the trained interviewer will then administer the baseline questionnaire in the participant's home.

The questionnaire will collect demographic data, as well as information on current dietary intake, drinking water treatment, knowledge of iron deficiency anemia, knowledge of malaria, and perceptions of supplement use.

Participants will have a venous blood sample taken at 0, 6, and 12 months and analyzed for hemoglobin and multiple biomarkers of iron status (e.g. soluble transferrin receptor, ferritin, and retinol binding protein (RBP)). Ferritin will be corrected for inflammation using measures of alpha-1 acid glycoprotein (AGP, g/L) and C-reactive protein (CRP, mg/L) which are biomarkers of chronic and acute inflammation, respectively.

Genotyping will be conducted to determine the prevalence of hemoglobinopathies among women. The prevalence of malaria in this cohort will be determined using rapid diagnostic test kits for P. Falciparum, and P. Vivax at baseline, midline, and endline.

Potential Significance: The LIF has the potential to be a low cost, effective and simple-to-use product to prevent and reduce iron deficiency anemia in Cambodia.

ELIGIBILITY:
Inclusion Criteria:

* Mild or Moderate Anemia [Hb 80-119]
* Willing to provide a fingerprick sample of blood at baseline
* Willing to provide 10 mL of venous blood at 0, 6 & 12 months
* Not planning on moving in the next 12 months
* Not participating in any other nutrition intervention
* Be able to provide written and information consent

Exclusion Criteria:

* Be ill or taking any medications [Hb < 80]
* Have normal Hb status [Hb > 120]
* Currently consuming or planning to consume Fe supplements in the next 12 months
* Pregnant (based on self report)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
hemoglobin concentration at endline | 12 months

SECONDARY OUTCOMES:
Change in ferritin concentration | Baseline (t=0), midline (t=6 months), and endline (t=12 months)
  Ferritin is a biomarker of iron status. Ferritin will be corrected with measures using measures of alpha-1 acid glycoprotein and C-reactive protein.
Number of women in Preah Vihear, Cambodia with a genetic hemoglobin disorder | Midline (t=6 months)
How the prevalence of malaria changes in women living in Preah Vihear Cambodia over one year | Baseline (t=0), midline (t=6 months), and endline (t=12 months)
Change in soluble transferrin receptor (sTfR) concentration | Baseline (t=0), midline (t=6 months), and endline (t=12 months)
  sTfR is a biomarker of iron status

CONTACTS AND LOCATIONS:
Overall Officials: Tim J Green, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Rovieng Health Centre, Rovieng Tboung, Preah Vihear, Cambodia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Rappaport AI, Whitfield KC, Chapman GE, Yada RY, Kheang KM, Louise J, Summerlee AJ, Armstrong GR, Green TJ. Randomized controlled trial assessing the efficacy of a reusable fish-shaped iron ingot to increase hemoglobin concentration in anemic, rural Cambodian women. Am J Clin Nutr. 2017 Aug;106(2):667-674. doi: 10.3945/ajcn.117.152785. Epub 2017 Jun 14. PMID 28615257